CLINICAL TRIAL: NCT07225790
Title: Emulation of the MONARCH-3 Trial Using Specialty Oncology Electronic Health Records Databases
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor, Brigham and Women's Hospital
Other Study IDs: 2022P002556-ENC-MONARCH-3; 75F40122C00181 (Other Grant/Funding Number: Food and Drug Administration)
Record Dates: First submitted 2025-11-05; First posted 2025-11-10 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Letrozole; Anastrozole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Initiation of abemaciclib plus letrozole/anastrozole: Any doses and frequency observed in clinical practice will be allowed
  Interventions: Drug: Initiation of abemaciclib plus letrozole/anastrozole
- Initiation of letrozole/anastrozole: Any doses and frequency observed in clinical practice will be allowed
  Interventions: Drug: Initiation of letrozole/anastrozole

INTERVENTIONS:
Drug: Initiation of abemaciclib plus letrozole/anastrozole — Any doses and frequency observed in clinical practice will be allowed
  Groups: Initiation of abemaciclib plus letrozole/anastrozole
Drug: Initiation of letrozole/anastrozole — Any doses and frequency observed in clinical practice will be allowed
  Groups: Initiation of letrozole/anastrozole

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale emulation of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
Randomized controlled trials (RCTs) are generally regarded as the gold-standard of evidence for establishing efficacy of medical products. However, real-world data (RWD) are increasingly used to complement evidence from RCTs. Yet, to have confidence in the accuracy of non-interventional studies medical products and their outcomes in oncology, investigators need to know what questions can be validly answered, with which non-interventional study designs, and which analysis methods are appropriate, given the data that is available. Building on a process from the RCT DUPLICATE initiative1-4 EmulatioN of Comparative Oncology trials with Real-world Evidence (ENCORE) is part of the expansion project specific to oncology and aims to emulate 12 randomized oncology RCTs using multiple EHR data sources.

The purpose of this protocol is to describe the emulation of the MONARCH-3 trial. MONARCH 3 is a double-blind, randomized phase III study of abemaciclib or placebo plus a nonsteroidal aromatase inhibitor in 493 postmenopausal women with hormone receptor (HR)-positive, human epidermal growth factor receptor 2 (HER2)-negative advanced breast cancer who had no prior systemic therapy in the advanced setting. Patients received abemaciclib or placebo (150 mg twice daily continuous schedule) plus either 1 mg anastrozole or 2.5 mg letrozole/anastrozole, daily.

ELIGIBILITY:
Inclusion Criteria:

* Female aged ≥18 years at treatment initiation from 2017 - 2023
* Evidence of metastatic breast cancer (MBC)
* Documentation of Estrogen/Progesterone receptor-positive (ER/PR+)
* Documentation of Human Epidermal Growth Factor Receptor Negative (HER2-)
* ECOG performance status of 0 or 1 within 90 days of index date

Exclusion Criteria:

* CNS metastases
* Prior treatment with CKD4/6 inhibitor
* Prior or current treatment with chemotherapy or endocrine therapy other than letrozole/anastrozole for systemic anticancer therapy for MBC.
* Prior (neo-)adjuvant endocrine therapy
* Systemic anticancer therapy other than abemaciclib or letrozole/anastrozole
* Non-breast cancer malignancy other than basal/squamous cell skin cancer or carcinoma in situ of cervix

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with ER/PR-positive, HER2-negative locally advanced or metastatic breast cancer who receive treatment without curative intent
Sampling Method: Non-Probability Sample
Enrollment: 3883 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Time to all-cause mortality (overall survival) | From time of initiation of therapy through the earliest of death from any cause (the primary outcome of interest) or end of data availability (depending on specialty oncology registry data provider, end of data ranges from June 2023 to April 2024)
  Hazard ratio (95% CI)

SECONDARY OUTCOMES:
Time to next treatment (TTNT) | From time of initiation of therapy through the earliest of TTNT, death from any cause, or end of data availability (depending on specialty oncology registry data provider, end of data ranges from June 2023 to April 2024)
  Hazard ratio (95% CI)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital; Denys Shay, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT07225790/Prot_SAP_001.pdf